CLINICAL TRIAL: NCT02384421
Title: Adaptive Closed Loop Neuromodulation and Neural Signatures of Parkinson's Disease
Acronym: aDBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Helen M. Bronte-Stewart, MD MSE, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 30880
Record Dates: First submitted 2015-02-18; First posted 2015-03-10 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Activa PC+S Neurostimulator (Experimental): Participants will be own controls and undergo both adaptive and continuous deep brain stimulation testing paradigms using Nexus D research tool
  PC+S: Primary Cell+Sensing
  Interventions: Device: Adaptive DBS (Activa PC+S Neurostimulator); Device: Continuous DBS (Activa PC+S Neurostimulator)

INTERVENTIONS:
Device: Adaptive DBS (Activa PC+S Neurostimulator)
  Other Names: Adaptive deep brain stimulation
Device: Continuous DBS (Activa PC+S Neurostimulator)
  Other Names: continuous deep brain stimulation

SUMMARY:
Continuous deep brain stimulation (cDBS) is an established therapy for the major motor signs in Parkinson's disease. Currently, cDBS is limited to "open-loop" stimulation, without real-time adjustment to the patient's state of activity, fluctuations and types of motor symptoms, medication dosages, or neural markers of the disease. The purpose of this study is to determine if an adaptive DBS system, responding to patient specific, clinically relevant neural or kinematic feedback, is efficacious on the motor Unified Parkinson's Disease Rating Scale (UPDRS III) and specific phenotypic measures in Parkinson's Disease compared to OFF therapy (i.e., OFF DBS and withdrawn from medication) and more efficient than cDBS. Not every recruited participant completed every part of the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of idiopathic Parkinson's disease, with bilateral symptoms at Hoehn and Yahr Stage greater than or equal to II.
2. Documented improvement in motor signs on versus off dopaminergic medication, with a change in the Unified Parkinson's Disease Rating Scale motor (UPDRS III) score of >= 30% off to on medication.
3. The presence of complications of medication such as wearing off signs, fluctuating responses and/or dyskinesias, and/or medication refractory tremor, and/or impairment in the quality of life on or off medication due to these factors.
4. Subjects should be on stable doses of medications, which should remain unchanged until the DBS system is activated. After the DBS system is optimized (during which time the overall medication dose may be reduced to avoid discomfort and complications such as dyskinesias) the medication dose should remain unchanged, if possible, for the duration of the study.
5. Treatment with carbidopa/levodopa, and with a dopamine agonist at the maximal tolerated doses as determined by a movement disorders neurologist.
6. Ability and willingness to return for study visits, at the initial programming and after three, six and twelve months of DBS.
7. Age > 18

Exclusion Criteria:

1. Subjects with significant cognitive impairment and/or dementia as determined by a standardized neuropsychological battery.
2. Subjects with clinically active depression, defined according to the Diagnostic and Statistical manual of Mental Disorders, Fourth Edition (DSM-IV) criteria and as scored on a validated depression assessment scale.
3. Subjects with very advanced Parkinson's disease, Hoehn and Yahr stage 5 on medication (non-ambulatory).
4. Age > 80.
5. Subjects with an implanted electronic device such as a neurostimulator, cardiac pacemaker/defibrillator or medication pump.
6. Subjects, who are pregnant, are capable of becoming pregnant, or who are breast feeding.
7. Patients with cortical atrophy out of proportion to age or focal brain lesions that could indicate a non-idiopathic movement disorder as determined by MRI
8. Subjects having a major comorbidity increasing the risk of surgery (prior stroke, severe hypertension, severe diabetes, or need for chronic anticoagulation other than aspirin).
9. Subjects having any prior intracranial surgery.
10. Subjects with a history of seizures.
11. Subjects, who are immunocompromised.
12. Subjects with an active infection.
13. Subjects, who require diathermy, electroconvulsive therapy (ECT), or transcranial magnetic stimulation (TMS) to treat a chronic condition.
14. Subjects, who have an inability to comply with study follow-up visits.
15. Subjects, who are unable to understand or sign the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-01; Primary Completion 2019-09-23 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Bronte-Stewart, MD MSE, Principal Investigator — Stanford University
Locations (1):
- Stanford Movement Disorders Center, Stanford, California, United States

REFERENCES:
- [Result] Velisar A, Syrkin-Nikolau J, Blumenfeld Z, Trager MH, Afzal MF, Prabhakar V, Bronte-Stewart H. Dual threshold neural closed loop deep brain stimulation in Parkinson disease patients. Brain Stimul. 2019 Jul-Aug;12(4):868-876. doi: 10.1016/j.brs.2019.02.020. Epub 2019 Feb 25. PMID 30833216
- [Result] Malekmohammadi M, Herron J, Velisar A, Blumenfeld Z, Trager MH, Chizeck HJ, Bronte-Stewart H. Kinematic Adaptive Deep Brain Stimulation for Resting Tremor in Parkinson's Disease. Mov Disord. 2016 Mar;31(3):426-8. doi: 10.1002/mds.26482. Epub 2016 Jan 27. No abstract available. PMID 26813875
- [Result] Petrucci MN, Neuville RS, Afzal MF, Velisar A, Anidi CM, Anderson RW, Parker JE, O'Day JJ, Wilkins KB, Bronte-Stewart HM. Neural closed-loop deep brain stimulation for freezing of gait. Brain Stimul. 2020 Sep-Oct;13(5):1320-1322. doi: 10.1016/j.brs.2020.06.018. Epub 2020 Jul 4. No abstract available. PMID 32634599

RESULTS

PARTICIPANT FLOW:
Groups:
- Activa PC+S Neurostimulator: Participants will be own controls and undergo both Adaptive DBS (Activa PC+S Neurostimulator) and Continuous DBS (Activa PC+S Neurostimulator) deep brain stimulation testing paradigms using Nexus D research tool
  PC+S: Primary Cell+Sensing
Period: Overall Study
Arm/Group | Activa PC+S Neurostimulator
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Activa PC+S Neurostimulator: Participants will be own controls and undergo both Adaptive DBS and Continuous DBS deep brain stimulation
Arm/Group | Activa PC+S Neurostimulator
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
Mean OFF UPDRS-III at Initial Programming [Mean (Standard Deviation); unit: UPDRS-III Score] — Scores on the UPDRS III range from 0-132. Higher scores represent a worse outcome.
  UPDRS-III Score | 41.9 (15.4)

OUTCOME MEASURES:

1. Primary Outcome: Normalized Beta Band Power (13-30 Hz) During aDBS
Description: Beta Band Power will be recorded continuously during intervention (30 minutes). The PC+S streams off power of the local field potential signal measured from the subthalamic nucleus in a frequency band of interest within the beta band (13-30 Hz). The amplitude of the signal, beta power, was streamed from each subthalamic nucleus (STN) during the calibration period of the experiment when DBS was off (i.e., OFF therapy), when continuous DBS was set at the lower and upper stimulation voltage that were found for determining the stimulation limits of adaptive DBS, and during the 30 minutes of aDBS. We calculated the median observed beta power during aDBS. To compute normalized beta band power, the median value was divided by the observed beta power OFF therapy and during the continuous DBS at the lower and upper voltage. A value less than 1 indicates reduced beta power during aDBS compared to the other conditions.
Time Frame: 30 minutes
Population: Participants who were assessed for this outcome and with no artifacts in the local field potential signal.
Measure: Mean (Standard Deviation); unit: Normalized median beta power
Units Other Than Participants: STNs
Arm/Group | Activa PC+S Neurostimulator
Number analyzed (Participants) | 13
Number analyzed (STNs) | 20
Normalized median beta power | 0.26 (0.14)
Statistical Analysis 1: Comparison: Activa PC+S Neurostimulator; Test type: Superiority; p < 0.001, t-test, 2 sided

2. Primary Outcome: Change in UPDRS III Score
Description: Movement Disorder Society's Unified Parkinson's Disease Rating Scale III (UPDRS III) score will be measured after 30 minutes of intervention and compared to baseline. Scores on the UPDRS III range from 0-132. Higher scores represent a worse outcome.
  For some participants, a modified UPDRS III was used in which items 3.9, 3.10, 3.11, 3.12, and 3.13 were excluded to only focus on the seated portion of the assessment, or only one hemibody was tested if the aDBS controller was only controlling one subthalamic nucleus.
Time Frame: 30 minutes
Population: Participants who were assessed for this outcome (had a clinical UPDRS assessment).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Activa PC+S Neurostimulator: Participants will be own controls and undergo both Adaptive and Continuous deep brain stimulation. OFF refers to off therapy (i.e. withdrawn medication and no deep brain stimulation). aDBS refers to an adaptive DBS based on a neural controller.
Arm/Group | Activa PC+S Neurostimulator
Number analyzed (Participants) | 8
score on a scale
  OFF | 28.1 (17.1)
  aDBS | 12.5 (10.5)
Statistical Analysis 1: Comparison: Activa PC+S Neurostimulator; Test type: Superiority; p = 0.0064, t-test, 2 sided

3. Secondary Outcome: Disease Symptoms (Tremor)
Description: Mean tremor power calculated from a triaxial gyroscope using a fast Fourier transform averaged between 4 and 8 Hz. Higher tremor power indicates worse tremor.
Time Frame: 30 minutes
Population: Participants who were assessed for this outcome and not excluded due to lack of tremor.
Measure: Mean (Standard Deviation); unit: (rad/s)^2
Units Other Than Participants: STNs
Groups:
- Activa PC+S Neurostimulator: Participants will be own controls and undergo both Adaptive and Continuous deep brain stimulation. OFF refers to off therapy (i.e. withdrawn medication and no deep brain stimulation). aDBS refers to an adaptive DBS based on a kinematic controller.
Arm/Group | Activa PC+S Neurostimulator
Number analyzed (Participants) | 5
Number analyzed (STNs) | 10
(rad/s)^2
  OFF | 0.040 (0.11)
  aDBS | 0.0072 (0.018)
Statistical Analysis 1: Comparison: Activa PC+S Neurostimulator; Test type: Superiority; p = 0.014, t-test, 2 sided

4. Secondary Outcome: Disease Symptoms (Freezing of Gait)
Description: Percent time freezing during a stepping-in-place task. Higher percent time freezing represents a worse outcome.
Time Frame: 30 minutes
Population: Participants who were assessed for this outcome and with no artifacts in the local field potential signal, artifacts in the kinematic data, or excluded since they did not identify as freezers.
Measure: Mean (Standard Deviation); unit: percentage of time freezing
Arm/Group | Activa PC+S Neurostimulator
Number analyzed (Participants) | 5
percentage of time freezing
  OFF | 22 (30)
  aDBS | 0 (1)
Statistical Analysis 1: Comparison: Activa PC+S Neurostimulator; Test type: Superiority; p = 0.25, Wilcoxon Signed-Rank Test

5. Secondary Outcome: Disease Symptoms (Bradykinesia)
Description: The root mean squared of the angular velocity during a wrist-flexion extension task. Higher root mean squared of angular velocity represents a better outcome.
Time Frame: 30 minutes
Population: Participants who were assessed for this outcome and with no artifacts in the local field potential signal, substantial tremor in the tested limb, or technical issues during the kinematic recording.
Measure: Mean (Standard Deviation); unit: root mean squared of angular velocity
Arm/Group | Activa PC+S Neurostimulator
Number analyzed (Participants) | 13
root mean squared of angular velocity
  OFF | 352.58 (56.46)
  aDBS | 457.44 (58.96)
Statistical Analysis 1: Comparison: Activa PC+S Neurostimulator; Test type: Superiority; p = 0.003, t-test, 2 sided

6. Secondary Outcome: DBS Voltage
Description: The median stimulation voltage during the aDBS run was determined for each individual's subthalamic nucleus. The overall group mean of the median stimulation voltages was compared to the group mean of the clinical continuous DBS (cDBS) median voltages.
Time Frame: 30 minutes
Population: Participants who were assessed for this outcome and with no artifacts in the local field potential signal.
Measure: Mean (Standard Deviation); unit: median stimulation voltage
Units Other Than Participants: STNs
Groups:
- Activa PC+S Neurostimulator: Participants will be own controls and undergo both Adaptive and Continuous deep brain stimulation. cDBS refers to Clinical Open Loop DBS. aDBS refers to an adaptive DBS based on a neural controller.
Arm/Group | Activa PC+S Neurostimulator
Number analyzed (Participants) | 13
Number analyzed (STNs) | 20
median stimulation voltage
  Clinical Open Loop (cDBS) | 3.12 (0.54)
  aDBS | 2.03 (0.91)
Statistical Analysis 1: Comparison: Activa PC+S Neurostimulator; Test type: Superiority; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to six years
Arm/Group | Activa PC+S Neurostimulator
All-Cause Mortality (participants affected / at risk) | 1/22
Serious Adverse Events (participants affected / at risk) | 4/22
Other Adverse Events (participants affected / at risk) | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Activa PC+S Neurostimulator (N=22)
Infection (Infections and infestations) | 1 (1) — serious, anticipated, device related
Lead/Connection Break (Product Issues) | 1 (1) — serious, anticipated, device related
Suicidality (Psychiatric disorders) | 1 (1) — serious, unanticipated, non-device related
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) — serious, unanticipated, non-device related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Activa PC+S Neurostimulator (N=22)
Device Failure (Product Issues) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Tenderness (Surgical and medical procedures) | 1 (1)
Sensing Malfunction (Product Issues) | 1 (1)
Device Malfunction (Product Issues) | 2 (2)
Gait Difficulties (Nervous system disorders) | 1 (1)
Speech (Nervous system disorders) | 1 (1)
Cognitive Difficulties (Nervous system disorders) | 1 (1)
Tingling (General disorders) | 4 (4)
Balance (General disorders) | 5 (6)
Muscle Soreness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle Contractions (Musculoskeletal and connective tissue disorders) | 10 (18)
Cognitive Problems (Nervous system disorders) | 5 (6)
Speech Difficulties (Nervous system disorders) | 13 (19)
Depression (Psychiatric disorders) | 3 (4)
Suicidal Ideation (Psychiatric disorders) | 1 (1)
Slowness (Musculoskeletal and connective tissue disorders) | 2 (3)
Stiffness (Musculoskeletal and connective tissue disorders) | 10 (16)
Walking Difficulty (Musculoskeletal and connective tissue disorders) | 16 (27)
Anxiety (Psychiatric disorders) | 3 (3)
Pain/Soreness (General disorders) | 4 (5)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Urinary Issues (Renal and urinary disorders) | 2 (2)
Weight changes (General disorders) | 5 (7)
Sleep Difficulties (Nervous system disorders) | 8 (12)
Weakness (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (15)
Hernia (Gastrointestinal disorders) | 1 (1)
Difficult Swallowing/Salivation (Gastrointestinal disorders) | 6 (7)
Stroke (Nervous system disorders) | 1 (1)
Mood (Psychiatric disorders) | 3 (3)
Dreaming (Nervous system disorders) | 1 (1)
Cough/Throat (Infections and infestations) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (2)
Dizziness (General disorders) | 2 (2)
Restless Leg (Nervous system disorders) | 2 (2)
Headache/Migraine (General disorders) | 2 (2)
Delerium (Psychiatric disorders) | 1 (1)
Vision problems (Eye disorders) | 4 (4)
Kidney Issues (Renal and urinary disorders) | 1 (1)
Blood Pressure (Cardiac disorders) | 1 (1)
Body Temperature (General disorders) | 3 (4)
Hair Loss (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT02384421/Prot_SAP_ICF_000.pdf